CLINICAL TRIAL: NCT01796002
Title: Phase 3 Multi-center Randomized Study to Compare Efficacy and Safety of Romidepsin CHOP (Ro-CHOP) Versus CHOP in Patients With Previously Untreated Peripheral T-cell Lymphoma
Brief Title: Efficacy and Safety of Romidepsin CHOP vs CHOP in Patients With Untreated Peripheral T-Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ro-CHOP Study
Record Dates: First submitted 2013-01-31; First posted 2013-02-21 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: PTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental: Romidepsin plus CHOP (Experimental): Patients in experimental arm receive romidepsin plus CHOP (Ro-CHOP) administered in 3 week cycles for 6 cycles.
  Romidepsin is administered at a dose of 12 mg/m² IV on day 1 and day 8 every 3 weeks.
  Interventions: Drug: Romidepsin + CHOP
- Standard: CHOP (Active Comparator): Patients in control Arm receive cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered in 3 week cycles for 6 cycles.
  Interventions: Drug: CHOP

INTERVENTIONS:
Drug: Romidepsin + CHOP — Ro-CHOP administered in 3 week cycles for 6 cycles or until progression Romidepsin is administered at a dose of 12 mg/m² IV on day 1 and day 8 every 3 weeks.
  Arms: Experimental: Romidepsin plus CHOP
Drug: CHOP — CHOP (cyclophosphamide, doxorubicin, vincristine and prednisone) administered in 3 week cycles for 6 cycles.
  Arms: Standard: CHOP

SUMMARY:
Primary objective of the study is to compare the efficacy of romidepsin when administered with CHOP versus CHOP alone in subjects with previously untreated peripheral T-cell lymphoma (PTCL) in terms of progression-free survival (PFS) assessed according to Response criteria for malignant lymphoma 1999 by a Response Adjudication Committee (RAC).

DETAILED DESCRIPTION:
This is a randomized multi-center phase III study, to compare efficacy and safety of Ro-CHOP with standard CHOP regimen in patients with previously untreated, histologically proven PTCL. Given the nature of the experimental agent, this study is an open-label study. Patients are randomized 1:1 to receive either (Arm A) cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) administered in 3 week cycles for 6 cycles [22] or (Arm B) romidepsin CHOP (Ro-CHOP) administered in 3 week cycles for 6 cycles. In the Ro-CHOP arm, romidepsin will be administered at a dose of 12 mg/m² IV on day 1 and day 8 every 3 weeks. In this study, patients will advance through three phases of the study: screening phase, treatment phase and follow-up phase. Patients will receive study drug(s) for up to 6 cycles, or until unacceptable toxicity will develop or progression or voluntary withdrawal. Patients will be followed for survival until the earliest of either 80% of patients have died or 3 years from the last patient randomized. Three years after the primary analysis an update of the database will be done and a rerun of the analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of 18 years of age to 80 years of age.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Patients with histologically proven peripheral T-cell lymphoma (PTCL), not previously treated; the following subtypes as defined by the World Health Organization (WHO) classification (2008;2011) may be included, whatever the Ann Arbor stage (I - IV):

   a. Nodal types: i. PTCL, not otherwise specified ii. Angioimmunoblastic T-cell lymphoma iii. Anaplastic large cell lymphoma, anaplastic lymphoma kinase (ALK)-negative type

   b. Extra-nodal types: i. Enteropathy-associated T-cell lymphoma ii. Hepato-splenic T-cell lymphoma iii. Subcutaneous panniculitis-like T-cell lymphoma iv. Primary cutaneous gamma-delta T-cell lymphoma v. Primary cutaneous cluster of differentiation 8 positive (CD8+) aggressive epidermotropic lymphoma vi. Primary cutaneous cluster of differentiation 4 positive (CD4+) small/medium T-cell lymphoma

   c. Other non classifiable peripheral T-cell lymphoma
5. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
6. Negative pregnancy test for Females of ChildBearing Potential (FCBP)
7. Female patients of child bearing potential must use an effective method of birth control (i.e. hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide or abstinence) during treatment period and 1 month thereafter; Males must use an effective method of birth control during treatment period and 3 months thereafter.
8. Life expectancy of ≥ 90 days (3 months).

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study.
2. Any condition that confounds the ability to interpret data from the study.
3. Other types of lymphomas, e.g. B-cell lymphoma
4. The following types of T cell lymphomas:

   1. Adult T-cell lymphoma/leukemia (HTLV-1 related T-cell lymphoma)
   2. Extranodal T-cell/Natural Killer (NK)-cell lymphoma, nasal type
   3. Anaplastic large cell lymphoma, ALK-positive type
   4. Cutaneous T cell lymphoma (mycosis fungoid, Sézary syndrome)
   5. Primary cutaneous cluster of differentiation antigen 30 positive (CD30+) T-cell lymphoproliferative disorder
   6. Primary cutaneous anaplastic T-cell lymphoma
5. Previous treatment for PTCL with immunotherapy or chemotherapy except for short-term corticosteroids (duration of ≤ 8 days) before randomization
6. Previous radiotherapy for PTCL except if localized to one lymph node area
7. Patients planned for autologous or allogeneic transplant as consolidation in first line
8. Central nervous system -meningeal involvement
9. Contraindication to any drug contained in the chemotherapy regimen,
10. Subjects with HIV positivity
11. Subjects with active hepatitis B or C. Chronic carriers of Hepatitis B virus (HBV) without HBV DNA positive blood are eligible. Subjects with non-active hepatitis C (with normal transaminases) are eligible.
12. Any of the following laboratory abnormalities, except if secondary to the lymphoma:

    1. Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L),
    2. Platelet count < 100,000/mm3 (100 x 109/L), or < 75,000/mm3 if bone marrow is involved,
    3. Serum Aspartate Aminotransferase (ASAT/AST) or Alanine Aminotransferase (ALAT/ALT) ≥ 3.0 x Upper Limit of Normal (ULN),
    4. Serum total bilirubin > 2 x ULN, except in case of hemolytic anemia,
    5. K+ and Mg2+ levels < Lower Limit of Normal (LLN), except if corrected per protocol guidance before beginning the romidepsin infusion
13. Serum creatinine > 2.0 x ULN
14. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast or untreated prostatic cancer without any plan for a treatment) unless the patient has been free of the disease for ≥ 3 years
15. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
16. Any known cardiac abnormalities such as:

    1. Patients with congenital long QT syndrome
    2. Corrected QT interval > 480 msec (using the Fridericia formula)
    3. Myocardial infarction within 6 months of cycle 1 day 1
    4. History of or concomitant significant cardiovascular disease
    5. Ejection fraction <45% by multigated acquisition (MUGA) scan or by echocardiogram;
17. Concomitant use of drugs that may cause a significant prolongation of the corrected QT interval (QTc)
18. Patients who have received more than 200 mg/m2 doxorubicin
19. Concomitant use of strong CYP3A4 inhibitors
20. Concomitant use of therapeutic warfarin due to a potential drug interaction. Use of a low dose of warfarin or another anticoagulant to maintain patency of venous access port and cannulas is permitted.
21. Clinically significant active infection
22. Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug
23. Pregnant or lactating females or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is Progression Free Survival | 60 months
  The primary efficacy endpoint is Progression Free Survival (PFS) using the response criteria for malignant lymphoma (1999) by a Response Adjudication Committee

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel BACHY, Professor, Study Chair — CH Lyon Sud, Pierre Bénite, France; Vincent CAMUS, MD, Study Chair — Centre Henri Becquerel, Rouen, France
Locations (131):
- Belgium (12):
  - ZNA Stuivenberg, Antwerp
  - A.Z. Sint Jan AV, Bruges
  - Institut Jules Bordet, Brussels
  - UCL Louvain Saint Luc, Brussels
  - ULB - Hôpital Erasme, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Hôpital Jolimont, Haine-Saint-Paul
  - AZ VUB, Jette
  - AZ Groeninge, Kortrijk
  - CHC - Clinique Saint Joseph, Liège
  - CHU de Liege, Liège
  - CHU Mont Godinne, Yvoir
- France (67):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH de Annecy, Annecy
  - CH Henri Duffaut, Avignon
  - CH Côte Basque, Bayonne
  - CHU Jean Minjoz, Besançon
  - CH de Béziers, Béziers
  - CHU de Bordeaux - Hôpital Haut Lévêque - Centre François Magendie, Bordeaux
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH du Dr Duchenne, Boulogne-sur-Mer
  - CH de Bourg en Bresse, Bourg-en-Bresse
  - Centre François Baclesse, Caen
  - Institut d'Hématologie de Basse-Normandie, Caen
  - CH de Chalon sur Saône, Chalon-sur-Saône
  - CH de Chambéry, Chambéry
  - Hôpital Antoine Béclère, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Pasteur, Colmar
  - CH Sud Francilien de Corbeil, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CH de Dunkerque, Dunkirk
  - CHU de Grenoble, Grenoble
  - CHD La Roche sur Yon, La Roche-sur-Yon
  - Centre Hospitalier de Versailles - André Mignot, Le Chesnay
  - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CH du Mans, Le Mans
  - Clinique Victor Hugo, Le Mans
  - CH de Lens, Lens
  - CHRU de Lille - Hôpital Claude Hurriez, Lille
  - CH de Saint Quentin, Lille
  - Hôpital Saint Vincent de Paul, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - CH de Saint Germain, Mantes-la-Jolie
  - Chi Poissy /Saint- Germain-En-Laye, Mantes-la-Jolie
  - Institut Paoli Calmettes, Marseille
  - CH de Meaux, Meaux
  - CHR de Metz, Metz
  - Hôpital Saint Eloi, Montpellier
  - CHU de Mulhouse, Mulhouse
  - CHU Nancy Brabois, Nancy
  - CHU Hôtel Dieu Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - CHU de Nîmes - Caremeau, Nîmes
  - Hôpital Necker, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Saint Louis, Paris
  - Institut Curie, Paris
  - CH de Perpignan, Perpignan
  - Centre François Magendie, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - CHU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - CH de Roubaix, Roubaix
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Centre René Huguenin, Saint-Cloud
  - CHU de Toulouse, Toulouse
  - CHU Bretonneau, Tours
  - CH Valence, Valence
  - CH de Valenciennes, Valenciennes
  - CH de Bretagne Atlantique, Vannes
  - Institut Gustave Roussy, Villejuif
- Germany (18):
  - Charité Medical School Campus Benjamin Franklin, Berlin
  - Charité Medical School Campus Virchow-Klinikum, Berlin
  - HELIOS Hospital Berlin-Buch, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Uniklinik Köln, Cologne
  - St Johannes-Hospital, Dortmund
  - Universitätsklinikum Carl Gustav Carus der TU Dresden, Dresden
  - Klinik Universitätsklinikum Düsseldorf, Düsseldorf
  - University of Duisburg-Essen, Essen
  - Krankenhaus Nordwest, Frankfurt am Main
  - Universitätklinikum Freiburg Klinik für Innere medizin I, Freiburg im Breisgau
  - UniversitätsKrebszentrum Göttingen - G-CCC, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikum St. Georg gGmbH, Leipzig
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Universitätsklinikum Ulm, Ulm
- Italy (10):
  - Istituto di Ematologia "Saragnoli" Policlinico San'Orsola-Malpighi, Bologna, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Ospedale Ferrarotto, Catania
  - Azienda Sanitaria Ospedaliera S.Croce e Carle Cuneo, Cuneo
  - Azienda Ospedaliera universitaria Careggi, Florence
  - Ematologia Oncologica Istituto Pascale, Napoli
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Ematologia Università La Sapienza, Roma
  - AOU San Giovanni Battista, Torino
  - Clinica Ematologica di Udine, Udine
- Instituto Português Oncologia, Lisbon, Portugal
- Singapore (3):
  - National Cancer Centre Singapore, Singapore
  - National University Cancer Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (6):
  - Dong-A Univ. Hospital, Busan
  - National Cancer Center, Goyang-si
  - Asian Medical Center, Seoul
  - Korean Cancer Center Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital Yonsei University, Seoul
- Spain (14):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - ICO l'Hospitalet, Barcelona
  - ICO - Institut Català d'Oncologia - Hospital Doctor Josep Trueta, Girona
  - Hospital de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario 12 de Octubre, Madrid
  - H. Morales Messeguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - H. Virgen del Rocío, Seville
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitario Dr. Peset de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camus V, Thieblemont C, Gaulard P, Cheminant M, Casasnovas RO, Ysebaert L, Damaj GL, Guidez S, Pica GM, Kim WS, Lim ST, Andre M, Gutierrez N, Penarrubia MJ, Staber PB, Trotman J, Huttmann A, Stefoni V, Tucci A, Fogarty P, Farhat H, Abraham J, Abarah W, Belmecheri F, Ribrag V, Delfau-Larue MH, Cottereau AS, Itti E, Li J, Delarue R, de Leval L, Morschhauser F, Bachy E. Romidepsin Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone Versus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Patients With Previously Untreated Peripheral T-Cell Lymphoma: Final Analysis of the Ro-CHOP Trial. J Clin Oncol. 2024 May 10;42(14):1612-1618. doi: 10.1200/JCO.23.01687. Epub 2024 Feb 16. PMID 38364196
- [Derived] Bachy E, Camus V, Thieblemont C, Sibon D, Casasnovas RO, Ysebaert L, Damaj G, Guidez S, Pica GM, Kim WS, Lim ST, Andre M, Garcia-Sancho AM, Penarrubia MJ, Staber PB, Trotman J, Huttmann A, Stefoni V, Re A, Gaulard P, Delfau-Larue MH, de Leval L, Meignan M, Li J, Morschhauser F, Delarue R. Romidepsin Plus CHOP Versus CHOP in Patients With Previously Untreated Peripheral T-Cell Lymphoma: Results of the Ro-CHOP Phase III Study (Conducted by LYSA). J Clin Oncol. 2022 Jan 20;40(3):242-251. doi: 10.1200/JCO.21.01815. Epub 2021 Nov 29. PMID 34843406
- See also: MedlinePlus related topics: Lymphoma — http://www.nlm.nih.gov/medlineplus/lymphoma.html
- See also: Drug Information available for: Romidepsin — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0128517077&QV1=ROMIDEPSIN